CLINICAL TRIAL: NCT00558519
Title: An Intergroup Phase II Clinical Trial for Adolescents and Young Adults With Untreated Acute Lymphoblastic Leukemia (ALL)
Brief Title: Combination Chemotherapy in Treating Young Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-10403; CALGB-10403; ECOG C10403; CDR0000574230 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Leukemia
Keywords: B-cell adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Mercaptopurine; Methotrexate; pegaspargase; Thioguanine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy, radiotherapy) (Experimental): Patients are given a series of leukemia treatments that are divided into several sequential courses and different chemotherapy combinations of treatment. Please see the "Detailed Description" section for more information.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: mercaptopurine
Drug: methotrexate
Drug: pegaspargase
Drug: thioguanine
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating young patients with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter study. The purpose of this study is to improve the outcome of adolescents and young adults with acute lymphoblastic leukemia (ALL). The objectives of the study are described below.

OBJECTIVES:

* To describe the outcomes (i.e., complete response rate, event-free survival, disease-free survival [DFS], and overall survival [OS]) of adolescents and young adults with newly diagnosed acute lymphoblastic leukemia (ALL) treated with a pediatric chemotherapy regimen by adult hematologists/oncologists at multiple sites.
* To explore the feasibility of extending the "pediatric approach" to adult patients up to 40 years of age.
* To estimate the DFS and OS of these patients.
* To describe the toxicities observed in these patients.
* To compare the outcomes of patients treated on this protocol with appropriate similar patients (by age and disease characteristics) treated by pediatric oncologists on protocol COG-AALL0232.
* To evaluate the adherence of adult hematologists/oncologists and their patients to a "pediatric" ALL treatment regimen and identify reasons for variances.
* To analyze and describe the outcomes of patients treated on this study according to pretreatment characteristics such as age, gender, white blood cell count, other hematologic parameters, blood chemistry, immunophenotype, cytogenetics and molecular genetic characteristics, and treatment variables such as treatment site (academic center or community), and protocol adherence.
* To analyze and describe the outcomes of patients treated on this study according to baseline psychosocial characteristics, demographics, and family support.

The courses of treatment for the research study are described below.

* Remission induction therapy: Patients receive intrathecal (IT) cytarabine on day 1; vincristine IV on days 1, 8, 15, and 22; prednisone IV or orally twice daily on days 1-28; daunorubicin hydrochloride IV on days 1, 8, 15, and 22; pegaspargase IV or intramuscularly (IM) on day 4 or 5 or 6; and IT methotrexate on days 8 and 29*. Patients undergo bone marrow aspirate (BMA) and biopsy on day 29 to assess induction response and minimal residual disease status. Patients with M1 marrow (< 1% lymphoblasts) proceed to remission consolidation therapy. Patients with M2 marrow (> 5% but < 25% lymphoblasts) proceed to extended remission induction therapy. Patients with M3 marrow are removed from protocol therapy.

NOTE: *Patients with CNS3 disease also receive IT methotrexate on days 15 and 22.

* Extended remission induction therapy: Patients receive prednisone IV or orally twice daily on days 1-14; vincristine IV on days 1 and 8; pegaspargase IM or IV on day 4 or 5 or 6; and daunorubicin hydrochloride IV on day 1. Patients undergo BMA and biopsy on day 15. Patients with M1 marrow proceed to remission consolidation therapy. Patients with M2 or M3 bone marrow are removed from protocol therapy.
* Remission consolidation therapy: Patients receive cyclophosphamide IV on days 1 and 29; cytarabine IV or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39; oral mercaptopurine on days 1-14 and 29-42; vincristine IV on days 15, 22, 43, and 50; pegaspargase IM or IV on days 15 and 43; and IT methotrexate on days 1, 8, 15*, and 22*. Once blood counts recover, patients proceed to interim maintenance therapy.

NOTE: *Patients with CNS3 disease do not receive IT methotrexate on days 15 and 22.

* Interim maintenance therapy: Patients receive vincristine IV and methotrexate (Capizzi methotrexate) IV on days 1, 11, 21, 31, and 41; pegaspargase IM or IV on days 2 and 22; and IT methotrexate on days 1 and 31. Once blood counts recover (ANC ≥ 750/mm^3 and platelet count ≥ 75,000/mm^3), patients proceed to delayed intensification therapy.
* Delayed intensification therapy: Patients receive vincristine IV on days 1, 8, 15, 43, and 50; dexamethasone IV or orally twice daily on days 1-7 and 15-21; doxorubicin hydrochloride IV on days 1, 8, and 15; pegaspargase IM or IV on day 4 or 5 or 6 AND day 43; cyclophosphamide IV on day 29; cytarabine IV or SC on days 29-32 and 36-39; oral thioguanine on days 29-42; and IT methotrexate on days 1, 29, and 36. Once blood counts recover, patients proceed to maintenance therapy.
* Maintenance therapy: Patients receive vincristine IV on days 1, 29, and 57; dexamethasone IV or orally twice daily on days 1-5, 29-33, and 57-61; mercaptopurine orally on days 1-84; IT methotrexate on day 1*; and oral methotrexate on days 8, 15, 22, 29**, 36, 43, 50, 57, 64, 71, and 78.

Treatment repeats every 12 weeks for 2 years from the start of interim maintenance (for female patients) or 3 years from the start of interim maintenance (for male patients).

NOTE: *IT methotrexate is also given on day 29 of the first 4 courses of maintenance therapy.

NOTE: **Oral methotrexate is held on day 29 of the first 4 courses of maintenance therapy (when IT methotrexate is given).

* Radiotherapy: During the first course of maintenance therapy, patients with testicular disease undergo concurrent radiotherapy to the testes 5 days a week for 2.5 weeks (total dose 2400 cGy given in 12 daily fractions); patients with CNS3 disease undergo concurrent cranial radiotherapy 5 days a week for 2 weeks (total dose of 1800 cGy given in 10 daily fractions); and patients with T-cell ALL undergo concurrent cranial radiotherapy (total dose of 2400 cGy given in 10 daily fractions) 5 days a week for 2 weeks.

Patients may complete surveys at the end of courses 1, 2, and 4, at the end of all protocol treatment, and at 6 and 18 months after the end of all protocol treatment.

After completion of study treatment, patients are followed every 1-3 months for 3 years and then every 6 months for 7 years.

ELIGIBILITY:
Eligibility Criteria:

1. Diagnosis

   1. Newly diagnosed patients with either B-precursor or T-precursor acute lymphoblastic leukemia (WHO criteria). Burkitt type leukemia as defined per protocol is not eligible. Patients known to have Ph+ ALL at time of diagnosis are not eligible.
   2. CALGB patients entered on CALGB 10403 who are later found to meet the following criteria for Ph+ ALL should have treatment on this trial discontinued and should be encouraged to enroll on CALGB 10001 or its successor trial:

      * BCR-ABL fusion transcript determined by FISH or RT-PCR
      * t(9;22)(q34;q11) or variant determined by cytogenetics

   Non-CALGB study participants who are later found to be Ph+ should have treatment on this trial discontinued and should be encouraged to enroll on an appropriate clinical trial specifically designed for Ph+ ALL.
2. Age: 16 - 39 years
3. ECOG Performance Status 0-2
4. Patients with Down Syndrome are excluded from this study due to the likelihood of excessive toxicity resulting. These patients should be treated in consultation with a pediatric oncologist.
5. Prior Therapy - No prior therapy except for limited treatment with corticosteroids or hydroxyurea and a single dose of intrathecal cytarabine.

   1. No prior therapy for acute leukemia except emergency therapy (corticosteroids or hydroxyurea) for blast cell crisis, superior vena cava syndrome, or renal failure due to leukemic infiltration of the kidneys. When indicated, leukapheresis or exchange transfusion is recommended to reduce the WBC.
   2. Single-dose intrathecal cytarabine is allowed prior to registration or prior to initiation of systemic therapy for patient convenience. This is usually done at the time of the diagnostic bone marrow or venous line placement to avoid a second lumbar puncture. Systemic chemotherapy must begin within 72 hours of this intrathecal therapy.
   3. Patients receiving prior steroid therapy are eligible for study. The dose and duration of previous steroid therapy should be carefully documented on case report forms.

Ages: 16 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 318 (Actual)
Dates: Start 2008-03-12 (Actual); Primary Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, M.D., Study Chair — University of Chicago

REFERENCES:
- [Background] Bleyer A: Older adolescents and young adults with acute lymphoblastic leukemia (ALL) in the United States: from the lowest to highest death rate and number of deaths--more rationale for the CALBG-SWOG-ECOG C10403 trial based on COG AALL0232. [Abstract] J Clin Oncol 26 (Suppl 15): A-18034, 2008.
- [Derived] Advani AS, Larsen E, Laumann K, Luger SM, Liedtke M, Devidas M, Chen Z, Yin J, Foster MC, Claxton D, Coffan K, Tallman MS, Appelbaum FR, Erba H, Stone RM, Hunger SP, McNeer JL, Loh ML, Raetz E, Winick N, Carroll W, Larson RA, Stock W. Comparison of CALGB 10403 (Alliance) and COG AALL0232 toxicity results in young adults with acute lymphoblastic leukemia. Blood Adv. 2021 Jan 26;5(2):504-512. doi: 10.1182/bloodadvances.2020002439. PMID 33496745
- [Derived] Stock W, Luger SM, Advani AS, Yin J, Harvey RC, Mullighan CG, Willman CL, Fulton N, Laumann KM, Malnassy G, Paietta E, Parker E, Geyer S, Mrozek K, Bloomfield CD, Sanford B, Marcucci G, Liedtke M, Claxton DF, Foster MC, Bogart JA, Grecula JC, Appelbaum FR, Erba H, Litzow MR, Tallman MS, Stone RM, Larson RA. A pediatric regimen for older adolescents and young adults with acute lymphoblastic leukemia: results of CALGB 10403. Blood. 2019 Apr 4;133(14):1548-1559. doi: 10.1182/blood-2018-10-881961. Epub 2019 Jan 18. PMID 30658992

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pediatric Regimen): Patients received induction (Course I), consolidation (Course II), interim maintenance (Course III), delayed intensification (Course IV), and long-term maintenance therapy (Course V). Please see the "Detailed Description" section for more information.
Period: Overall Study
Arm/Group | Treatment (Pediatric Regimen)
Started | 318
Completed | 295
Not Completed | 23
Not completed — Ph+ | 20
Not completed — Ineligible | 1
Not completed — Insufficient data | 1
Not completed — Never received treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pediatric Regimen)
Number analyzed (Participants) | 295
Age, Continuous [Median (Full Range); unit: years] | 24.0 [17.0 to 39.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 180

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Complete response rate is defined as the percentage of patients who achieve bone marrow response (defined using the M bone marrow criteria for acute lymphoblastic leukemia (ALL); if M0 to M1 status (blast cells ,5%) was achieved by the end of induction or extended induction, the patient was considered a responder) at the end of induction therapy.
Time Frame: Up to 8 years post-registration
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Pediatric Regimen)
Number analyzed (Participants) | 295
percentage of patients | 89 [85 to 92]

2. Primary Outcome: Event-free Survival
Description: EFS was defined as time from registration in this study to the earliest occurrence of any of the following: failure to achieve bone marrow response (defined using the M bone marrow criteria for acute lymphoblastic leukemia (ALL); if M0 to M1 status (blast cells ,5%) was achieved by the end of induction or extended induction, the patient was considered a responder) by day 60, death, relapse at any site, or development of second malignant disease.
Time Frame: Up to 8 years post-registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pediatric Regimen)
Number analyzed (Participants) | 295
months | 78.1 [41.8 to NA] — The 95% confidence interval upper limit was not estimable (below the level of detection).

3. Primary Outcome: Disease-free Survival
Description: DFS was defined as time from bone marrow response in this study to the earliest occurrence of any of the following: failure to achieve bone marrow response (defined using the M bone marrow criteria for acute lymphoblastic leukemia (ALL); if M0 to M1 status (blast cells ,5%) was achieved by the end of induction or extended induction, the patient was considered a responder) by day 60, death, relapse at any site, or development of second malignant disease.
Time Frame: Up to 8 years post-registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pediatric Regimen)
Number analyzed (Participants) | 295
months | 81.7 [58.4 to NA] — The 95% confidence interval upper limit was not estimable (below the level of detection).

4. Primary Outcome: Overall Survival
Description: OS was defined from registration to death resulting from any cause.
Time Frame: Up to 8 years post-registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pediatric Regimen)
Number analyzed (Participants) | 295
months | NA [NA to NA] — The median and 95% confidence interval were not estimable (insufficient number of events/below the level of detection).

5. Primary Outcome: Number of Participants Who Experienced at Least One Grade 3 or Higher Adverse Event at Least Possibly Related to Treatment (Toxicity)
Description: The number of participants who experienced toxicity (defined as at least one grade 3 or higher adverse event at least possibly related to treatment) is reported below.
Time Frame: Up to 10 years post-registration
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pediatric Regimen)
Number analyzed (Participants) | 295
Participants | 286

6. Other Pre Specified Outcome: Analysis and Description of the Outcomes of Patients Treated on This Study According to Baseline Psychosocial Characteristics, Demographics, and Family Support
Time Frame: Up to 10 years post-registration
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Outcomes of Patients Treated on This Study According to Pretreatment Characteristics Such as Age, Gender, White Blood Cell Count, Other Hematologic Parameters, Blood Chemistry, Immunophenotype, Cytogenetics and Molecular Genetic Characteristics
Time Frame: Up to 10 years post-registration
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Adherence of Adult Hematologists/Oncologists and Their Patients to a "Pediatric" Acute Lymphoblastic Leukemia Treatment Regimen and Identification of Reasons for Variances
Time Frame: Up to 10 years post-registration
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Outcomes of Adolescent and Young Adult Patients Treated on This Study Compared With Those of Patients Treated Per COG-AALL0232
Time Frame: Up to 10 years post-registration
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment (Pediatric Regimen)
All-Cause Mortality (participants affected / at risk) | 105/295
Serious Adverse Events (participants affected / at risk) | 134/295
Other Adverse Events (participants affected / at risk) | 268/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pediatric Regimen) (N=295)
Blood disorder (Blood and lymphatic system disorders) | 4 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 67 (84)
Hemoglobin decreased (Blood and lymphatic system disorders) | 128 (209)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (4)
Atrial flutter (Cardiac disorders) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Cardiac disorder (Cardiac disorders) | 1 (1)
Cardiac pain (Cardiac disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 4 (5)
Pericardial effusion (Cardiac disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 30 (44)
Supraventricular tachycardia (Cardiac disorders) | 4 (6)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 4 (4)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 6 (6)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 5 (6)
Dry eye syndrome (Eye disorders) | 2 (2)
Extraocular muscle paresis (Eye disorders) | 2 (2)
Eye disorder (Eye disorders) | 4 (4)
Eye pain (Eye disorders) | 4 (5)
Flashing vision (Eye disorders) | 2 (2)
Optic nerve edema (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 2 (2)
Retinopathy (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 13 (14)
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 44 (57)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 6 (8)
Colonic hemorrhage (Gastrointestinal disorders) | 4 (4)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 39 (46)
Diarrhea (Gastrointestinal disorders) | 49 (63)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 20 (22)
Dysphagia (Gastrointestinal disorders) | 6 (7)
Esophageal mucositis (clin exam) (Gastrointestinal disorders) | 1 (1)
Esophageal mucositis (funct/sympt) (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 5 (5)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 4 (5)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 30 (33)
Nausea (Gastrointestinal disorders) | 95 (135)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 12 (12)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 13 (13)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 4 (4)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 4 (4)
Typhlitis (Gastrointestinal disorders) | 4 (4)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 64 (84)
Chest pain (General disorders) | 12 (13)
Chills (General disorders) | 30 (34)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 26 (31)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 87 (127)
Fever (General disorders) | 28 (38)
Flu-like symptoms (General disorders) | 1 (1)
Gait abnormal (General disorders) | 4 (4)
General symptom (General disorders) | 6 (8)
Ill-defined disorder (General disorders) | 4 (4)
Injection site reaction (General disorders) | 2 (4)
Localized edema (General disorders) | 14 (16)
Multi-organ failure (General disorders) | 1 (1)
Pain (General disorders) | 29 (41)
Bile duct stenosis (Hepatobiliary disorders) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 7 (7)
Hepatobiliary disease (Hepatobiliary disorders) | 5 (5)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 22 (25)
Immune system disorder (Immune system disorders) | 2 (2)
Colitis, infectious (Infections and infestations) | 4 (4)
Opportunistic infection (Infections and infestations) | 1 (1)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 63 (77)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 9 (13)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Intraop. inj. - Appendix (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Activated partial throm time prolonged (Investigations) | 35 (42)
Alanine aminotransferase increased (Investigations) | 125 (198)
Alkaline phosphatase increased (Investigations) | 56 (81)
Amylase increased (Investigations) | 14 (16)
Aspartate aminotransferase increased (Investigations) | 116 (187)
Blood bilirubin increased (Investigations) | 99 (138)
Blood prolactin abnormal (Investigations) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Coagulopathy (Investigations) | 4 (5)
Creatine phosphokinase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 33 (38)
Electrocardiogram QTc interval prolonged (Investigations) | 2 (2)
Fibrinogen decreased (Investigations) | 73 (100)
Gamma-glutamyltransferase increased (Investigations) | 9 (10)
INR increased (Investigations) | 19 (24)
Laboratory test abnormal (Investigations) | 16 (19)
Leukocyte count decreased (Investigations) | 66 (99)
Lipase increased (Investigations) | 20 (22)
Lymphocyte count decreased (Investigations) | 45 (65)
Neutrophil count decreased (Investigations) | 126 (201)
Platelet count decreased (Investigations) | 126 (197)
Serum cholesterol increased (Investigations) | 15 (19)
Weight gain (Investigations) | 7 (8)
Weight loss (Investigations) | 18 (19)
Acidosis (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 36 (46)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 8 (11)
Blood glucose increased (Metabolism and nutrition disorders) | 111 (170)
Blood uric acid increased (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 12 (12)
Glucose intolerance (Metabolism and nutrition disorders) | 7 (7)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Renal tubular disorder (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 69 (94)
Serum calcium decreased (Metabolism and nutrition disorders) | 61 (85)
Serum calcium increased (Metabolism and nutrition disorders) | 7 (7)
Serum glucose decreased (Metabolism and nutrition disorders) | 30 (38)
Serum magnesium decreased (Metabolism and nutrition disorders) | 35 (49)
Serum magnesium increased (Metabolism and nutrition disorders) | 27 (27)
Serum phosphate decreased (Metabolism and nutrition disorders) | 20 (22)
Serum potassium decreased (Metabolism and nutrition disorders) | 59 (81)
Serum potassium increased (Metabolism and nutrition disorders) | 20 (21)
Serum sodium decreased (Metabolism and nutrition disorders) | 62 (90)
Serum sodium increased (Metabolism and nutrition disorders) | 11 (14)
Serum triglycerides increased (Metabolism and nutrition disorders) | 24 (33)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (49)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 10 (12)
Joint disorder (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (10)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 12 (14)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (19)
Myositis (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (11)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 17 (18)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 35 (40)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Accessory nerve disorder (Nervous system disorders) | 1 (1)
Arachnoiditis (Nervous system disorders) | 2 (3)
Ataxia (Nervous system disorders) | 2 (3)
Central nervous system necrosis (Nervous system disorders) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 3 (3)
Depressed level of consciousness (Nervous system disorders) | 5 (7)
Dizziness (Nervous system disorders) | 36 (47)
Dysgeusia (Nervous system disorders) | 9 (9)
Encephalopathy (Nervous system disorders) | 2 (2)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 86 (118)
Hypoglossal nerve disorder (Nervous system disorders) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2)
Leukoencephalopathy (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 4 (4)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 8 (10)
Oculomotor nerve disorder (Nervous system disorders) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 14 (20)
Peripheral sensory neuropathy (Nervous system disorders) | 68 (97)
Seizure (Nervous system disorders) | 10 (10)
Speech disorder (Nervous system disorders) | 7 (7)
Syncope (Nervous system disorders) | 4 (5)
Tremor (Nervous system disorders) | 5 (5)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 22 (27)
Confusion (Psychiatric disorders) | 9 (9)
Depression (Psychiatric disorders) | 26 (32)
Euphoria (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 41 (45)
Libido decreased (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 5 (6)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (2)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Kidney pain (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 8 (8)
Urethral pain (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Urine discoloration (Renal and urinary disorders) | 5 (5)
Urogenital disorder (Renal and urinary disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 9 (10)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (38)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30 (34)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngeal mucositis (clin exam) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (22)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Hand-and-foot syndrome/reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 8 (9)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (7)
Rash desquamating (Skin and subcutaneous tissue disorders) | 26 (31)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 6 (6)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 6 (6)
Sweating (Skin and subcutaneous tissue disorders) | 15 (15)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (5)
Flushing (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 6 (6)
Hemorrhage (Vascular disorders) | 3 (4)
Hypertension (Vascular disorders) | 10 (12)
Hypotension (Vascular disorders) | 21 (23)
Thrombosis (Vascular disorders) | 23 (26)
Vascular disorder (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pediatric Regimen) (N=295)
Blood disorder (Blood and lymphatic system disorders) | 10 (10)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 13 (14)
Febrile neutropenia (Blood and lymphatic system disorders) | 114 (181)
Hemoglobin decreased (Blood and lymphatic system disorders) | 259 (1235)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Lymphatic disorder (Blood and lymphatic system disorders) | 5 (5)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 7 (7)
Cardiac disorder (Cardiac disorders) | 6 (7)
Cardiac pain (Cardiac disorders) | 2 (2)
Edema (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 22 (29)
Pericardial effusion (Cardiac disorders) | 8 (8)
Pericarditis (Cardiac disorders) | 2 (2)
Premature ventricular contractions (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 9 (10)
Sinus tachycardia (Cardiac disorders) | 66 (120)
Supraventricular tachycardia (Cardiac disorders) | 6 (7)
Ventricular bigeminy (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 8 (13)
Ear disorder (Ear and labyrinth disorders) | 9 (9)
Ear pain (Ear and labyrinth disorders) | 16 (19)
External ear inflammation (Ear and labyrinth disorders) | 2 (2)
External ear pain (Ear and labyrinth disorders) | 7 (7)
Hearing impaired (Ear and labyrinth disorders) | 5 (7)
Middle ear inflammation (Ear and labyrinth disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 7 (7)
Cushingoid (Endocrine disorders) | 14 (28)
Endocrine disorder (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (4)
Diplopia (Eye disorders) | 4 (4)
Dry eye syndrome (Eye disorders) | 9 (11)
Extraocular muscle paresis (Eye disorders) | 7 (9)
Eye disorder (Eye disorders) | 28 (36)
Eye pain (Eye disorders) | 9 (9)
Eyelid function disorder (Eye disorders) | 2 (3)
Flashing vision (Eye disorders) | 4 (4)
Photophobia (Eye disorders) | 14 (15)
Retinopathy (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 43 (57)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 32 (35)
Abdominal pain (Gastrointestinal disorders) | 105 (185)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 5 (10)
Colitis (Gastrointestinal disorders) | 9 (9)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 141 (290)
Diarrhea (Gastrointestinal disorders) | 127 (257)
Dry mouth (Gastrointestinal disorders) | 13 (24)
Dyspepsia (Gastrointestinal disorders) | 64 (113)
Dysphagia (Gastrointestinal disorders) | 13 (15)
Enteritis (Gastrointestinal disorders) | 1 (1)
Esophageal mucositis (clin exam) (Gastrointestinal disorders) | 1 (1)
Esophageal mucositis (funct/sympt) (Gastrointestinal disorders) | 3 (3)
Esophageal pain (Gastrointestinal disorders) | 7 (7)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 6 (8)
Flatulence (Gastrointestinal disorders) | 12 (13)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 13 (15)
Gastrointestinal disorder (Gastrointestinal disorders) | 35 (82)
Gingival pain (Gastrointestinal disorders) | 10 (11)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 17 (22)
Ileus (Gastrointestinal disorders) | 3 (3)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3)
Malabsorption (Gastrointestinal disorders) | 2 (2)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 86 (133)
Nausea (Gastrointestinal disorders) | 221 (724)
Oral hemorrhage (Gastrointestinal disorders) | 14 (18)
Oral pain (Gastrointestinal disorders) | 22 (24)
Pancreatitis (Gastrointestinal disorders) | 24 (30)
Periodontal disease (Gastrointestinal disorders) | 2 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 15 (23)
Rectal mucositis (clin exam) (Gastrointestinal disorders) | 1 (1)
Rectal mucositis (funct/sympt) (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 8 (8)
Rectal ulcer (Gastrointestinal disorders) | 1 (1)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1)
Salivary gland fistula (Gastrointestinal disorders) | 1 (1)
Small intestinal mucositis (funct/sympt) (Gastrointestinal disorders) | 1 (1)
Small intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 16 (20)
Tooth development disorder (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 6 (14)
Toothache (Gastrointestinal disorders) | 15 (18)
Typhlitis (Gastrointestinal disorders) | 4 (4)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 172 (405)
Chest pain (General disorders) | 40 (53)
Chills (General disorders) | 56 (77)
Edema limbs (General disorders) | 83 (149)
Facial pain (General disorders) | 6 (6)
Fatigue (General disorders) | 214 (733)
Fever (General disorders) | 80 (110)
Flu-like symptoms (General disorders) | 12 (12)
Gait abnormal (General disorders) | 4 (4)
General symptom (General disorders) | 22 (29)
Hypothermia (General disorders) | 1 (1)
Ill-defined disorder (General disorders) | 4 (5)
Injection site reaction (General disorders) | 7 (8)
Localized edema (General disorders) | 28 (45)
Pain (General disorders) | 68 (106)
Visceral edema (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 6 (6)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 7 (14)
Cytokine release syndrome (Immune system disorders) | 6 (10)
Hypersensitivity (Immune system disorders) | 34 (37)
Immune system disorder (Immune system disorders) | 5 (8)
Serum sickness (Immune system disorders) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Colitis, infectious (Infections and infestations) | 11 (15)
Conjunctivitis (Infections and infestations) | 1 (2)
Opportunistic infection (Infections and infestations) | 3 (3)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 161 (265)
Viral hepatitis (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 39 (62)
Device complication (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative complications (Injury, poisoning and procedural complications) | 1 (1)
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 4 (4)
ADH abnormal (Investigations) | 1 (1)
Activated partial throm time prolonged (Investigations) | 69 (179)
Alanine aminotransferase increased (Investigations) | 247 (1359)
Alkaline phosphatase increased (Investigations) | 117 (308)
Amylase increased (Investigations) | 25 (29)
Aspartate aminotransferase increased (Investigations) | 240 (1107)
Blood bilirubin increased (Investigations) | 206 (673)
CD4 lymphocytes decreased (Investigations) | 2 (6)
Coagulopathy (Investigations) | 11 (14)
Creatine phosphokinase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 71 (101)
Electrocardiogram QTc interval prolonged (Investigations) | 4 (4)
Fibrinogen decreased (Investigations) | 166 (289)
Gamma-glutamyltransferase increased (Investigations) | 22 (59)
Haptoglobin decreased (Investigations) | 1 (2)
INR increased (Investigations) | 49 (112)
Laboratory test abnormal (Investigations) | 33 (74)
Leukocyte count decreased (Investigations) | 162 (793)
Lipase increased (Investigations) | 45 (60)
Lymphocyte count decreased (Investigations) | 116 (600)
Neutrophil count decreased (Investigations) | 256 (1240)
Platelet count decreased (Investigations) | 255 (1151)
Serum cholesterol increased (Investigations) | 20 (41)
Weight gain (Investigations) | 27 (61)
Weight loss (Investigations) | 57 (95)
Acidosis (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 117 (237)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 16 (36)
Blood glucose increased (Metabolism and nutrition disorders) | 232 (1019)
Blood uric acid increased (Metabolism and nutrition disorders) | 29 (55)
Dehydration (Metabolism and nutrition disorders) | 37 (45)
Glucose intolerance (Metabolism and nutrition disorders) | 4 (4)
Iron overload (Metabolism and nutrition disorders) | 3 (6)
Obesity (Metabolism and nutrition disorders) | 2 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 142 (344)
Serum calcium decreased (Metabolism and nutrition disorders) | 129 (311)
Serum calcium increased (Metabolism and nutrition disorders) | 14 (21)
Serum glucose decreased (Metabolism and nutrition disorders) | 65 (125)
Serum magnesium decreased (Metabolism and nutrition disorders) | 61 (123)
Serum magnesium increased (Metabolism and nutrition disorders) | 34 (45)
Serum phosphate decreased (Metabolism and nutrition disorders) | 50 (75)
Serum potassium decreased (Metabolism and nutrition disorders) | 130 (267)
Serum potassium increased (Metabolism and nutrition disorders) | 40 (48)
Serum sodium decreased (Metabolism and nutrition disorders) | 136 (296)
Serum sodium increased (Metabolism and nutrition disorders) | 23 (37)
Serum triglycerides increased (Metabolism and nutrition disorders) | 31 (58)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 14 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 82 (188)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 127 (297)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 17 (22)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 4 (7)
Joint range motion decr cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 53 (98)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 35 (55)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 68 (162)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 33 (48)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 76 (96)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 9 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 104 (224)
Slipped femoral epiphysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (1)
Arachnoiditis (Nervous system disorders) | 2 (2)
Ataxia (Nervous system disorders) | 4 (4)
Cerebrospinal fluid leakage (Nervous system disorders) | 8 (8)
Cognitive disturbance (Nervous system disorders) | 7 (7)
Depressed level of consciousness (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 89 (169)
Dysgeusia (Nervous system disorders) | 34 (46)
Extrapyramidal disorder (Nervous system disorders) | 4 (4)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 199 (607)
Intracranial hemorrhage (Nervous system disorders) | 6 (6)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2)
Leukoencephalopathy (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 12 (29)
Mini mental status examination abnormal (Nervous system disorders) | 3 (3)
Neuralgia (Nervous system disorders) | 7 (13)
Neurological disorder NOS (Nervous system disorders) | 21 (23)
Peripheral motor neuropathy (Nervous system disorders) | 35 (84)
Peripheral sensory neuropathy (Nervous system disorders) | 202 (891)
Seizure (Nervous system disorders) | 9 (11)
Speech disorder (Nervous system disorders) | 5 (6)
Syncope (Nervous system disorders) | 6 (6)
Syncope vasovagal (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 16 (25)
Agitation (Psychiatric disorders) | 11 (15)
Anxiety (Psychiatric disorders) | 98 (194)
Confusion (Psychiatric disorders) | 13 (14)
Depression (Psychiatric disorders) | 76 (168)
Euphoria (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 123 (236)
Libido decreased (Psychiatric disorders) | 4 (5)
Personality change (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 6 (6)
Bladder hemorrhage (Renal and urinary disorders) | 3 (3)
Bladder pain (Renal and urinary disorders) | 3 (3)
Bladder spasm (Renal and urinary disorders) | 2 (3)
Cystitis (Renal and urinary disorders) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 6 (6)
Kidney pain (Renal and urinary disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1)
Urethral pain (Renal and urinary disorders) | 3 (3)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 23 (31)
Urinary incontinence (Renal and urinary disorders) | 9 (15)
Urinary retention (Renal and urinary disorders) | 8 (11)
Urine discoloration (Renal and urinary disorders) | 9 (9)
Urogenital disorder (Renal and urinary disorders) | 20 (33)
Breast pain (Reproductive system and breast disorders) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 5 (6)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 5 (6)
Ovarian hemorrhage (Reproductive system and breast disorders) | 1 (2)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 4 (6)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 4 (5)
Testicular pain (Reproductive system and breast disorders) | 2 (2)
Uterine hemorrhage (Reproductive system and breast disorders) | 2 (6)
Uterine pain (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 20 (25)
Vaginal pain (Reproductive system and breast disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 59 (93)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 116 (256)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 87 (172)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 50 (67)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 15 (21)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Laryngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal mucositis (clin exam) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (clin exam) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pharyngeal mucositis (funct/sympt) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 46 (64)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 28 (42)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Tracheal mucositis (funct/sympt) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 75 (155)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 6 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 17 (22)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 (5)
Hand-and-foot syndrome/reaction (Skin and subcutaneous tissue disorders) | 8 (11)
Nail disorder (Skin and subcutaneous tissue disorders) | 7 (13)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 24 (32)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 38 (48)
Rash acneiform (Skin and subcutaneous tissue disorders) | 30 (56)
Rash desquamating (Skin and subcutaneous tissue disorders) | 95 (180)
Scalp pain (Skin and subcutaneous tissue disorders) | 2 (3)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 37 (68)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (4)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 4 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 11 (14)
Sweating (Skin and subcutaneous tissue disorders) | 57 (91)
Urticaria (Skin and subcutaneous tissue disorders) | 9 (9)
Flushing (Vascular disorders) | 6 (7)
Hematoma (Vascular disorders) | 13 (16)
Hemorrhage (Vascular disorders) | 14 (15)
Hot flashes (Vascular disorders) | 15 (23)
Hypertension (Vascular disorders) | 38 (82)
Hypotension (Vascular disorders) | 55 (75)
Lymphedema (Vascular disorders) | 2 (3)
Phlebitis (Vascular disorders) | 3 (4)
Thrombosis (Vascular disorders) | 43 (53)
Vascular disorder (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes